CLINICAL TRIAL: NCT04121702
Title: Outpatient Cardiac Tele-Rehabilitation in a Public Sports Center Versus Traditional Hospital Model
Brief Title: Outpatient Cardiac Tele-Rehabilitation in a Public Sports Center
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Juan Izquierdo García (Other)
Responsible Party: Sponsor-Investigator, Juan Izquierdo García, Juan Izquierdo García, Physical Therapist, Principal Investigator, Hospital Universitario 12 de Octubre
Organization: Hospital Universitario 12 de Octubre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: e-CARCEX
Record Dates: First submitted 2019-06-17; First posted 2019-10-10 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Acute Coronary Syndrome; Cardiac Rehabilitation; Telerehabilitation; Secondary Prevention; Wearable Electronic Devices; Exercise Therapy
Keywords: Cardiac Rehabilitation; Telerehabilitation; Secondary Prevention; Wearable Electronic Devices; Exercise Therapy
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEP-H (Active Comparator): Physical exercise program at a hospital
  Interventions: Procedure: Cardiac Rehabilitation
- PEP-PSC (Experimental): Physical exercise program with tele-monitoring in a public sport centre
  Interventions: Procedure: Cardiac Rehabilitation

INTERVENTIONS:
Procedure: Cardiac Rehabilitation — Implementation of a physical exercise program (PEP) with tele-monitoring

SUMMARY:
The aim of this study is to establish an innovative Cardiac Tele-Rehabilitation (CTR) model. It could expands assistance resources through coordination with public administrations, developing a physical exercise program (PEP) assistance model in phase II that resolves the current situation of lack of adherence in the PEP due in part to the long waiting time to start it. To sum up this study could improve adherence in Cardiac Rehabilitation Phase III. It represents an opportunity to validate an innovative model for the realization of the PEP for phase II that could be expanded to other centres.

DETAILED DESCRIPTION:
Cardiac Rehabilitation (CR) programs show benefits in cardiovascular morbidity and mortality, exercise capacity, risk factors and quality of life. The use of new information and communication technologies (ICT) allows remote monitoring of activity and rhythm, defining a new model of cardiac tele-rehabilitation (CTR) and proving to be safe.

The investigators intend to evaluate a new model of CR in Phase II in acute coronary syndrome (ACS), based on the implementation of the physical exercise program (PEP) in a public sports centre (PSC) with tele-monitoring by means of a wearable electronic device, S-PATCH3-Cardio, to compare the adherence of a PEP based on a CTR-PSC model with the traditional in-hospital program (PEP-H) maintaining the efficacy and safety of the CR program.

Patients with recent stratified ACS of low and / or moderate risk will be included who will be randomly assigned to the PEP-H group who will perform 18 PEP sessions with strength training and cardiorespiratory resistance in a hospital, or a CTR-PSC group that performs the 18 sessions of the PEP with strength training and cardiorespiratory resistance in the PSC.

All patients will perform the rest of the CR program at the hospital that it includes: functional tests, consultations with nurse, cardiologist, rehabilitation doctor, and the educational program, with 10 Workshops in a Cardio-healthy Classroom.

ELIGIBILITY:
Inclusion Criteria:

* Recent ACS (1-12 months) of low / moderate risk for the realization of a PEP and without physical impediments for it
* Availability of a mobile phone with Android operating system where you can install the S-PATCH3-Cardio application
* Patients who recognize that they are trained to operate the S-PATCH3-Cardio device after being instructed in its operation and perform a 24-hour simulation.
* Signature of informed consent

Exclusion Criteria:

* Baseline ergospirometry that does not reach maximalist criteria (respiratory quotient> 1.1)
* Mental disability
* Associated comorbidity that prevents performing PEP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-05-08 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Adherence to physical exercise | At the end of the program (6 weeks)
  Adherence to physical exercise measured by number of physical exercise sessions realized by each patient
Functional capacity | At the end of the program (6 weeks)
  Change of functional capacity measured by cardiopulmonary exercise test

SECONDARY OUTCOMES:
Glucose levels | At the end of the program (6 weeks)
  Evaluate changes on the glucose metabolic profile (mg/dL)
Glycated hemoglobin levels (HbA1c) | At the end of the program (6 weeks)
  Evaluate changes on the glycated hemoglobin (mg/dL)
Low-density lipoprotein (LDL) levels | At the end of the program (6 weeks)
  Evaluate changes on the LDL metabolic profile (mg/dL)
High-density lipoprotein (HDL) levels | At the end of the program (6 weeks)
  Evaluate changes on the HDL metabolic profile (mg/dL)
Total colesterol levels | At the end of the program (6 weeks)
  Evaluate changes on the total colesterol metabolic profile (mg/dL)
Blood pressure levels | At the end of the program (6 weeks)
  Evaluate changes on systolic and diastolic blood pressure levels (mmHg)
Smoking | At the end of the program (6 weeks)
  Evaluate changes on smoking status (cessation of smoking)
Weight | At the end of the program (6 weeks)
  Evaluate changes on weight (kg)
Abdominal perimeter | At the end of the program (6 weeks)
  Evaluate changes on abdominal perimeter (cm)
Body Mass Index (BMI) | At the end of the program (6 weeks)
  Evaluate changes on body mass index (weight in kg and height in meters will be combined to calculate BMI in kg/m˄2)
Adherence to Mediterranean Diet | At the end of the program (6 weeks)
  Evaluate changes on mediterranean dietary habits measured ussing the Mediterranean Diet Assessment Scale (MEDAS) which is constituted by 14 ítems with questions concerning dietary habits related to the medditerranean dietary style. Minimum score: 0, maximum score: 14. Values over 9 are corresponded to good adherence to mediterranean diet, values under 9 are considered to be bad adherence.
Phisical exercise profile | At the end of the program (6 weeks)
  Evaluate changes on level of physical activity measured ussing the International Physical Activity Questionnaire (IPAQ). It asks about three specific types of activity undertaken in the four domains: leisure time physical activity, domestic and gardening (yard) activities, work-related physical activity, transport-related physical activity. The specific types of activity that are assessed are walking, moderate-intensity activities and vigorous-intensity activities. Computation of the total score for the form requires summation of the duration (in minutes) and frequency (days) of walking, moderate-intensity and vigorous-intensity activities.
  Maximun value: the sum total of all Walking, Moderate and Vigorous time variables greater than 960 minutes (16 hours).
  Mínimum value: Only values of 10 or more minutes of activity should be included in the calculation of summary scores. Responses of less than 10 minutes [and their associated days] should be re-coded to 'zero'

CONTACTS AND LOCATIONS:
Overall Officials: Juan Izquierdo Garcia, Therapist, Principal Investigator — Hospital Universitario 12 de Octubre
Locations (1):
- Hospital Universitario 12 de Octubre, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No